CLINICAL TRIAL: NCT05639621
Title: Management of Meaningful Accompaniment as a Nursing Strategy to Reduce Patient Anxiety in Endoscopic Procedures in a Public Hospital, Year 2021: Randomized Clinical Trial.
Brief Title: Management of Meaningful Accompaniment to Reduce Patient Anxiety in Endoscopic Procedures: Randomized Clinical Trial
Acronym: MMEANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Concepcion (Other)
Responsible Party: Principal Investigator, Patricia Jara Concha, Dr, Full Professor, Universidad de Concepcion
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: University of Concepcion
Record Dates: First submitted 2021-10-16; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Anxiety State
Keywords: Significant accompaniment; anxiety; nursing; endoscopy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meaningful accompaniment (Experimental): Patient who is going to undergo an endoscopic procedure and who will have a significant accompaniment by a person freely chosen by the patient and who will escort him in a visual and tactile way during the pre-procedure, intra-procedure, and post-procedure endoscopic stage.
  Interventions: Procedure: Accompaniment
- Usual care (No Intervention): Patient who is going to undergo an endoscopic procedure and who receives regular care provided by the service during the pre-procedure, intra-procedure and post-procedure stage.

INTERVENTIONS:
Procedure: Accompaniment — presence of a person freely chosen by the patient, who will escort in a visual and tactile way during the endoscopic procedure
  Arms: Meaningful accompaniment

SUMMARY:
An upper digestive endoscopy diagnostic procedure is undoubtedly a situation that will generate anxiety. The environment, protocols, distance the patient from the family member or partner, which is perceived as a threat to integrity. The objective of the study is to determine the effectiveness of a structured, significant follow-up nursing intervention to reduce anxiety in patients who are going to undergo upper digestive endoscopy in a public hospital in the Biobío Region, year 2021. The methodological proposal will be in a randomized, single-blind, third-party evaluation clinical trial, the intervention will consist of the visual and tactile presence of a significant companion throughout the endoscopic procedure. The sample will be 126 that will make up the experimental and control group. It is hypothesized that patients who have a significant follow-up will obtain 10 points less on the anxiety scale compared to those who did not have the intervention. The data will be collected with the Spielberg state / anxiety test (STAIT) and the Visual Analog Scale (VAS) to measure psychological effects, with vital parameters (pressure, pulse, respiration, saturometry), physiological effects, as well as the effects biochemicals with blood levels of potassium, glycemia and cortisol in saliva and mechanical effects through the monitoring of movements, using a mesh of pressure sensors. The difference-in-difference statistical method will be applied by t student, to analyze the data. The requirements of Emmanuel will be applied to safeguard the ethics of the study. It is hoped that significant follow-up as a nursing intervention will be shown to reduce the anxiety of the patient who is going to undergo an endoscopic procedure.

DETAILED DESCRIPTION:
The study is a clinical trial, with random assignment to two groups: control and experimental, that is, the study corresponds to a Design with Pretest-Postest and Control Group. The sample will be made up of all the patients who will undergo an endoscopy procedure in a public hospital, during the first quarter of the year 2021 and the intervention will be the significant accompaniment that the patient who is going to undergo an endoscopic procedure of the group will have experimental (EG) in the pre-procedure stage - during the procedure and after the procedure, while the control group (CG) will receive the usual care of the service under study, that is, without a significant companion.

DESCRIPTION OF THE STAGES OF THE INTERVENTION

1. - PRE PROCEDURE PERIOD

   1. Mediate: Due to the COVID-19 pandemic contingency, it is necessary to adopt the necessary security measures before, during and after conducting the interview with the patient who is going to undergo an endoscopic procedure. In this context, in the mediate preoperative period, to inform the patient that he is going to undergo an endoscopic procedure, non-face-to-face interviews will be promoted, through the use of electronic means, through videoconferencing, recorded telephone calls or emails, if the patient so requires, as well as conducting face-to-face interviews according to the protocols provided for it. The selected patients will be contacted by the coordinating nurse 3 or 4 days in advance, informing them that they must approach the emergency service to take PCR test (to detect COVID-19, this telephone contact will be the one that the responsible researcher will use to propose the voluntary participation in the study. If approved, the nursing professional responsible for the study will request the signing of the informed consent on the day the patient and companion attend to take the PCR test.

      PROTOCOL SIGNATURE INFORMED CONSENT NOT PRESENTIAL

      To carry out this procedure, the following protocol will be followed with each of the patients and significant companions that will make up the study sample:
      1. Patient identification by name.
      2. Identification of the responsible researcher.
      3. Presentation of the research project.
      4. Request to approve recording of informed consent and / or sociodemographic data.
      5. Reading informed consent
      6. Request for clarification of doubts.
      7. Completion of the interview and acknowledgments.

      PROTOCOL SIGNATURE INFORMED CONSENT IN PERSON To carry out this procedure, the following protocol will be followed with each of the patients and significant companions that will make up the study sample.
      1. The interview will be carried out in an individual and well ventilated room.
      2. The following should be considered in the interview:

         * Avoid physical contact when greeting and maintain a social distance of 1 meter between the responsible researcher and the patient interviewed.
         * Hand hygiene with soap and water and / or alcohol gel solution after interview.
         * Use of personal protection elements (PPE): Use a surgical type mask that covers the nose and mouth, replace the mask each time it gets wet - dispose of the mask once removed in a garbage can with a lid.
      3. Patient identification by name
      4. Identification of the responsible researcher
      5. Presentation of the research project
      6. Request to approve recording of informed consent and / or sociodemographic data
      7. Reading informed consent and request for sociodemographic data (Annex 4)
      8. Request for clarification of doubts
      9. End of interview and acknowledgments
      10. Hand hygiene with soap and water and / or alcohol gel solution after the interview

      10) Cleaning of the place where the meeting was held after it was concluded 11) Keep the names, identification and telephone numbers of the interviewee for at least one month

      INTERVIEW ROOM CLEANING AND DISINFECTION PROCEDURE Before carrying out the disinfection of the interview room, a surface cleaning process must be carried out, by removing organic and inorganic matter, usually by friction, with the help of detergents used in the establishment under study, subsequently rinsing with water to eliminate dirt by dragging.

      Once the cleaning process has been carried out, the already clean surfaces must be disinfected, with the application of disinfectant products used by the service under study through the use of sprinklers, towels, fiber or microfiber cloths or mops.
   2. Inmediate: the day of the endoscopic procedure, the significant person will be received by the clinical nurse, who will be in charge of:

      * Give general and specific instructions on the procedure.
      * Hand hygiene with soap and water.
      * Delivery of costumes to enter at endoscopic procedure room. The significant companion will be next to the patient in the pre-procedure room and both will be accompanied by the nursing professional in charge of managing this monitoring, who will measure the patient the following parameters: Psychological, physiological, biochemical parameters.
2. - INTRAPROCEDURE PERIOD. Once the patient is on the endoscopic procedure table, the significant companion follows the instructions of the nursing professional, who leaves it on the patient's right side, takes the patient's hand for the duration of the sedation procedure. In this stage, after sedation, the responsible endoscopy medical professional will be asked for authorization to apply the Anxiety Assessment Scale (VAS), after which the investigated patient is asked to indicate the intensity of the sensation by placing a line at across the line, representing the intensity of the sensation at that moment. Once the patient is under sedation, the significant companion follows the instructions of the nursing professional, who tells to leave and accompanies the way to the waiting room.
3. - POSTPROCEDURE PERIOD. After sedation recovery, the nursing professional supervises the hygiene of the significant companion's hands, then leaves at the side of the patient's unit, will take the patient's hand until he regains consciousness. The nursing professional will measure the psychological-physiological-biochemical parameters. In this last stage, a variable that measures mechanical parameters will be incorporated, that is, the respiratory and body movements that the patient has in the post-sedation stage.

INTERVENTION IN CONTROL GROUP WILL CONSIST OF THE FOLLOWING STAGES:

I.- Preprocedure Period

1. Mediate Preoperative: In this context COVID-19, in the mediate preoperative period, to inform the patient that he is going to undergo a surgical procedure, non-face-to-face interviews will be promoted, through the use of electronic means, through videoconferencing, recorded telephone calls or e-mails, if the patient requires it, as well as conducting face-to-face interviews according to the protocols provided for it. The protocol for signing informed consent not in person and in person will be carried out in both groups.
2. Immediate: On the day of the endoscopic procedure, the patient will be accompanied by the nursing professional in charge of managing this monitoring, who will measure the following parameters: Psychological, physiological, biochemical parameters.

II.- Intraprocedure period After sedation, authorization will be requested from the responsible endoscopy medical professional to apply the Anxiety Assessment Scale (VAS), before which the investigated patient is asked to indicate the intensity of the sensation by placing a line through of the scale, which represents the intensity of anxiety at that moment.

III.- Postprocedure Period Once the patient has recovered from sedation, the evaluator will measure the psychological -physiological-biochemical parameters.

In this last stage, a variable that measures mechanical parameters will be incorporated, that is, the respiratory and body movements that the post-sedation patient has.

SAMPLE SIZE CALCULATION The statistical program Epidat 3.1 was used to calculate the sample size of the study. To carry out this procedure, the estimates from other studies were used, with a standard deviation of 10.4 for the STAY scale, with a difference of 5 points as clinically relevant. The level of significance was set at 0.05 (5%), a ratio between the means of 1, with a power of 80%. After entering the data into the software, the finally suggested sample is 126 patients, a number that is weighted to admit 10% of dropouts or withdrawals from the study, completing a sample size to be selected of 139 patients. From the definitive sample size (n = 126), the experimental group (n = 63) and the control group (n= 63) were finally formed.

DESCRIPTIVE ANALYSIS The data obtained will be analyzed through the SPSS statistical program. For the analysis of the data obtained, a statistical evaluation will be carried out by objectives, which will include, firstly, descriptive analysis through frequency tables and graphs, and secondly, obtaining statistics such as mean, standard deviation, coefficient of variation, maximum and minimum.

INFERENTIAL ANALYSIS FOR THE TEST OF HYPOTHESIS. For the development of this experimental study (intervention in a treatment group and counterfactual in a control group), the difference-in-difference method will be used, by means of the T-Student test. In this case, the comparisons are of three types.

First, the means of the control and experimental groups are compared in the baseline period, where it is expected that there are no significant differences. With this evaluation it is hoped to prove that both groups are homogeneous prior to the intervention.

Secondly, within each group, the means obtained in different periods (Preprocedure, Intraprocedure and Postprocedure) are compared, expecting that the control and experimental groups present a different behavior, in particular, that the eventual increases in the anxiety-related variables are lower in the experimental group compared to the control group.

Third, the means for the Preprocedure-Intraprocedure and Postprocedure periods are compared between the control and experimental groups, where better results are expected in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients who can read and write
* Patient who is the first endoscopy to undergo
* Patient who in previous hospitalizations have had no incidents.
* Patient participating throughout the surgical stage with a significant companion.
* Spanish speaking patients.
* Patients living in the Bío-Bío Region.
* Patients who have signed informed consent and agreed to participate voluntarily

Exclusion Criteria:

* Patients older than 85 years.
* Patients with psychiatric disorders.
* Patients with severe sensory alterations or disabilities that make the interview difficult.
* Patients with alterations or injuries in the hands that hinder sensitivity.
* Patients with treatments with sedatives and / or NSAIDs, since their use could affect blood pressure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Decrease 5 points on the anxiety scale. The preferred format is to use outcome-neutral language in Outcome Measure Title and Description (e.g., "change" instead of "decrease"). Please review and revise as appropriate. | 60 minutes measured before and after endoscopic procedure
  Patients who have a significant accompaniment structured follow-up have less 5 points on the anxiety scale compared to patients who did not have the intervention, with 0 points until 60 points and higher scores indicate a worse result.

SECONDARY OUTCOMES:
Mantainance or not increase of Psychological parameters | 30 minutes measured during the endoscopic procedure
  The Visual Analogue Scale will be used, with 0 points until 10 points and higher scores indicate a worse result.
Maintenance or not increase of physiological parameters | 60 minutes measured three times (before, during and after endoscopic procedure)
  Blood pressure, heart rate and saturometry are baseline parameters therefore its maintenance or not increase is the best result.
Maintenance or not increase of Biochemical parameters | 60 minutes measured two times (before and after endoscopic procedure)
  Blood and salivary cortisol levels and blood potassium and glucose levels are baseline parameters therefore its maintenance or not increase is the best result.

OTHER OUTCOMES:
Maintenance o not increase of mechanical parameters | 60 minutes (after endoscopic procedure)
  Breathing and body movements are baseline parameters therefore its maintenance or not increase is the best result.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Rodríguez, Study Director — Universidad de Concepcion
Locations (1):
- Hospital de Tome, Tomé, Concepcion, Chile